CLINICAL TRIAL: NCT03166267
Title: A Prospective Case Series Study to Monitor Healing Progression and Real Life Weight Bearing After Tibial Fracture Using Smart Biofeedback Systems
Brief Title: Real Life Weight Bearing After Tibial Fractures
Status: Completed | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: SmartFix II - Moticon
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2020-10

CONDITIONS: Tibial Fractures; External Fixation Pin Site Infection
MeSH Terms: conditions — Tibial Fractures | interventions — External Fixators

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: External fixator — Tibia fracture (AO 41-43) treated with external fracture fixation (large external fixator)

SUMMARY:
In this prospective case series patients with a tibial fracture are monitored with smart biofeedback systems to document the healing progression and real life weight.

DETAILED DESCRIPTION:
Ten patients treated with a large external fixator after tibial fracture will be enrolled for this prospective case series.

Patients will be equipped with the AO Fracture Monitor (a data logger device) attached post-operatively to a connection rod of the external fixator. The device continuously measures deformation of the fixator frame due to normal weight bearing for up to 12 months by means of a strain gauge. The strain signal is processed on-board and several parameters related to the loading characteristics of the fracture are stored.

Simultaneously, patients will be equipped with a fully integrated sensor insole (OpenGo Insole, Moticon GmbH, München). This product offers long-term weight bearing data (recording and storage) and allows non-invasive documentation of real life loading in patients without affecting the daily life activity of the patient. Recording of weight-bearing data will be obtained for a maximum of 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of tibial fracture (AO 41-43)
* External fracture fixation with large external fixator
* Capable of at least partial weight-bearing
* Bone segment transport (if applicable) must be completed
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/ Informed Consent Form (ICF)
  * Willingness and ability to participate in the clinical investigation according to the Clinical Investigation Plan (CIP)
  * Signed and dated Ethics Committee (EC)

Exclusion Criteria:

* External fixation as temporary stabilization
* Bone fragment compression
* Joint-bridging external fixation
* Any not medically managed severe systemic disease
* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the study period
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients from the participating clinic are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Loading patterns | Up to 4 months
  Average peak force per step

SECONDARY OUTCOMES:
Activity | Up to 4 months
  Patient activity measured as number of loading events per day
Healing | Up to 4 months
  Expert opinion
Pain level | Up to 4 months
  Numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Döbele, MD, Principal Investigator — BGU Tübingen
Locations (1):
- BGU Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No